CLINICAL TRIAL: NCT02211469
Title: A Randomized, Placebo-Controlled, Double-Blind, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986104 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM001-001
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 1-amino-3-((R)-6-hexyl-5,6,7,8-tetrahydronaphthalen-2-yl)cyclopentyl)methanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel 1: BMS-986104 or Placebo (Experimental): BMS-986104 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986104; Drug: Placebo
- Panel 2: BMS-986104 or Placebo (Experimental): BMS-986104 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986104; Drug: Placebo
- Panel 3: BMS-986104 or Placebo (Experimental): BMS-986104 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986104; Drug: Placebo
- Panel 4: BMS-986104 or Placebo (Experimental): BMS-986104 or Placebo single dose by mouth as specified
  Interventions: Drug: BMS-986104; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986104
Drug: Placebo

SUMMARY:
The primary objective in this study is to assess if single doses of BMS-986104 that are safe, tolerable, and result in sufficient lymphopenia (50% to 70% reduction in absolute lymphocyte count) can be achieved without bradycardia or other adverse events in healthy male subjects.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Healthy male subjects as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations will be eligible to participate in the study
* Men ages 18 to 49 years, inclusive

Exclusion Criteria:

* Any acute or chronic medical illness judged to be clinically-significant by the Investigator and/or Sponsor medical monitor
* Presence of fecal occult blood at screening
* History of prolonged occupational exposure to organic solvents or pesticides
* History of vitamin B12 deficiency and/or achlorhydria; or a vitamin B12 level at screening <lower limit of normal (LLN), confirmed by repeat test
* History of Guillain-Barré Syndrome
* Past or current history of central or peripheral neuropathies, or past or current symptoms of sustained or recurrent paresthesias (tingling), numbness, or neuropathic pain (burning, aching or stabbing) in any extremities. Note: Experiencing an extremity "falling asleep" occasionally is not be exclusionary
* Clinically significant abnormality in the neurological exam at baseline (predose)
* Clinically significant nerve electrophysiology abnormalities at baseline (predose)
* Any history of testicular or epididymal disease/disorder
* Clinically significant abnormality on ophthalmologic exam or any findings suggesting an increased risk of macular edema at baseline (predose)
* History of hypothyroidism or carpal tunnel syndrome
* Subjects with history of diabetes mellitus
* Subjects with history of any type of heart disease, including ischemia, infarction, arrhythmias, hypertension, atrioventricular block of any degree, bradycardia, syncope, clinically significant ECG abnormalities, or any congenital heart disease
* Subjects with any acute or chronic bacterial, fungal or viral infection within the last 3 months prior to screening, as well as any febrile illness of unknown origin within 14 days of screening
* Subjects who have received any live vaccines within 1 month of study drug administration or who plan to have a live vaccine at any time during the study
* Positive test for tuberculosis at screening (QuantiFERON® GOLD)

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events (AEs) / serious adverse events (SAEs) | Up to 1 month post discharge
Mean difference in ECG heart rate (HR) nadir values | Up to 4 days postdose
Nadir absolute lymphocyte count (ALC) defined as the lowest ALC measured at any time after the dose | Up to 4 days postdose

SECONDARY OUTCOMES:
Safety and tolerability based on severity, investigator causality assessment and outcomes of all AEs (regardless of seriousness criteria), association between AEs and study drug exposure parameters, and physical examination | Up to 1 month post discharge
Mean difference in ECG HR values in BMS-986104-treated versus placebo-treated healthy male subjects, identifying nadir ECG HR | Day -1 up to 24h and Days 1-5
Percent reduction in ECG HR | Day -1 up to 24h and Days 1-5
Time to nadir ECG HR | Day -1 up to 24h and Days 1-5
Maximum observed blood concentration (Cmax) of BMS-986104 | Up to Day 56
Time of maximum observed blood concentration (Tmax) of BMS-986104 | Up to Day 56
Terminal half-life (T-HALF) of BMS-986104 | Up to Day 56
Area under the blood concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of BMS-986104 | Up to Day 56
Area under the blood concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986104 | Up to Day 56
Apparent total clearance (CLT/F) of BMS-986104 | Up to Day 56
Apparent volume of distribution of terminal phase (Vz/F) of BMS-986104 | Up to Day 56
Metabolite to parent AUC(INF) ratio [MR_AUC(INF)] for both BMS-986104 and BMT-019434 | Up to Day 56
Effects of single oral doses of BMS-986104 on the following ALC | Up to 4 days postdose
  * Time to nadir ALC from time 0h (predose)
  * Percent reduction in ALC from baseline to nadir

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx